CLINICAL TRIAL: NCT03503292
Title: Using Pharmacogenomics (PGx) Results to Guide Post-operative Nausea and Vomiting (PONV) Treatment Practices: A Pilot Study
Brief Title: Pharmacogenomics and Post-Operative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yvette N. Martin, MD-PhD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-011283
Record Dates: First submitted 2018-04-03; First posted 2018-04-19 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Nausea
Keywords: Pharmacogenetics; CYP2D6; Ondansetron; Granisetron; Bariatric surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Granisetron; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYP2D6 rapid metabolizer (Experimental): Participants with CYP2D6 rapid metabolizer status will received granisetron for for post operative nausea and vomiting prophylaxis and treatment
  Interventions: Drug: Granisetron
- CYP2D6 normal metabolizer (Experimental): Participants with CYP2D6 poor or normal metabolizer status will received 4mg ondansetron for post operative nausea and vomiting prophylaxis and treatment
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Granisetron — Rapid metabolizer will receive 1mg IV Granisetron
  Other Names: Kytril
  Arms: CYP2D6 rapid metabolizer
Drug: Ondansetron — Poor or normal metabolizers will receive 4mg Ondansetron IV
  Other Names: Zofran
  Arms: CYP2D6 normal metabolizer

SUMMARY:
The Researchers overall goal is to evaluate the benefit and utility of preemptive genotypic data to guide post-operative nausea and vomiting treatment in the bariatric surgical population. The hypothesis is that using genotypic variation in CYP2D6 to select the appropriate 5HT3 serotonin receptor antagonist to treat PONV will decrease rates of PONV in the bariatric surgical population.

ELIGIBILITY:
Inclusion Criteria

* A Mayo Clinic patient scheduled to undergo any bariatric surgical procedure, including Roux-en-Y gastric bypass, sleeve gastrectomy, or duodenal switch.
* Patient age 18 or above.
* Patients must understand and provide written informed consent and HIPAA authorization prior to initiation of any study-specific procedures.
* Patient is willing to engage in a medication adjustment as part of their clinical visit (when needed).

Exclusion Criteria

* Patient with uncontrolled concurrent illness including psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent.
* Patients that deny access to their medical records for research purposes will not be included in this study. Also any patient who will be unable to have genetic testing at minimum of 1 week prior to scheduled surgery or with allergies to ondansetron or granisetron.
* Any patient with prior genetic testing that is readily available in the medical record will be excluded from this study.
* Any patient that is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette N Martin, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- CYP2D6 Rapid Metabolizer (Granisetron): Participants with CYP2D6 rapid metabolizer status received granisetron for for post operative nausea and vomiting prophylaxis and treatment
  Granisetron: Rapid metabolizer received 1mg IV Granisetron
- CYP2D6 Normal Metabolizer (Ondansetron): Participants with CYP2D6 poor or normal metabolizer status received 4mg ondansetron for post operative nausea and vomiting prophylaxis and treatment
  Ondansetron: Poor or normal metabolizers received 4mg Ondansetron IV
Period: Overall Study
Arm/Group | CYP2D6 Rapid Metabolizer (Granisetron) | CYP2D6 Normal Metabolizer (Ondansetron)
Started | 2 | 90
Completed | 2 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP2D6 Rapid Metabolizer (Granisetron) | CYP2D6 Normal Metabolizer (Ondansetron) | Total
Number analyzed (Participants) | 2 | 90 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (21.2) | 47.1 (13.0) | 47.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 78 | 80
  Male | 0 | 12 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 2 | 84 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 90 | 92
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 46.6 (15.9) | 45.4 (9.0) | 45.4 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Episodes of Postoperative Nausea
Description: The total number count of post operative nausea episodes were determined by nursing documentation or by treatment with rescue antinausea medication.
Time Frame: 0-48 hours post bariatric surgery
Measure: Number; unit: episodes
Arm/Group | CYP2D6 Rapid Metabolizer (Granisetron) | CYP2D6 Normal Metabolizer (Ondansetron)
Number analyzed (Participants) | 2 | 90
episodes | 0 | 16

2. Primary Outcome: Episodes of Postoperative Vomiting
Description: The total number count of post operative vomiting episodes were determined by nursing documentation or by treatment with rescue antinausea medication.
Time Frame: 0-48 hours post bariatric surgery
Measure: Number; unit: episodes
Arm/Group | CYP2D6 Rapid Metabolizer (Granisetron) | CYP2D6 Normal Metabolizer (Ondansetron)
Number analyzed (Participants) | 2 | 90
episodes | 0 | 4

ADVERSE EVENTS:
Time Frame: Adverse Events were collect from baseline (surgery) to one week post surgery, for approximately one week.
Arm/Group | CYP2D6 Rapid Metabolizer (Granisetron) | CYP2D6 Normal Metabolizer (Ondansetron)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/90
Other Adverse Events (participants affected / at risk) | 0/2 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03503292/Prot_SAP_000.pdf